CLINICAL TRIAL: NCT00905034
Title: Phase II Study of Methotrexate, Vincristine, Pegylated L-asparaginase and Dexamethasone (MOAD) in Acute Lymphoblastic Leukemia (ALL) Salvage
Brief Title: Methotrexate, Vincristine, Pegylated L-Asparaginase and Dexamethasone (MOAD) in Acute Lymphoblastic Leukemia (ALL) Salvage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Leadiant Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0267; NCI-2010-01147 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Leukemia, Lymphocytic, Acute
Keywords: Acute lymphoblastic leukemia; ALL; Leukemia; Methotrexate; Vincristine; PEG-l-asparaginase; PEG asparaginase; Pegaspargase; Oncaspar; Polyethylene Glycol Conjugated Lasparaginase-H; Dexamethasone; Decadron; Rituximab; Rituxan
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Methotrexate; Vincristine; pegaspargase; Dexamethasone; Calcium Dobesilate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MOAD (Experimental): Chemotherapy regimen of methotrexate, rituximab, vincristine, pegylated L-asparaginase and dexamethasone (MOAD).
  Interventions: Drug: Methotrexate; Drug: Vincristine; Drug: PEG-l-asparaginase; Drug: Dexamethasone; Drug: Rituximab

INTERVENTIONS:
Drug: Methotrexate — 200 mg/m^2 by vein on days 1 and 15.
  Other Names: Rheumatrex
Drug: Vincristine — 1.4 mg/m^2 by vein (maximum dose 2 mg) on days 1, 8 and 15.
  Other Names: Oncovin®
Drug: PEG-l-asparaginase — 2500 International units/m^2 by vein on days 2 and 16
  Other Names: Oncaspar®; PEG asparaginase; Pegaspargase; Polyethylene Glycol Conjugated Lasparaginase-H
Drug: Dexamethasone — 40 mg by vein or by mouth daily days 1-4 and 15-18.
  Other Names: Decadron®
Drug: Rituximab — Rituximab 375 mg/m^2 by vein on days 1 and 15 (first 4 cycles) for patients CD20 positive or positive by immunostain.
  Other Names: Rituxan®

SUMMARY:
This goal of this clinical research study is to learn if the combination of methotrexate, pegylated-L-asparaginase, vincristine, and dexamethasone (also rituximab in some patients) can help to control ALL that has not responded to previous treatment or has come back after a response or chronic myeloid leukemia (CML).

DETAILED DESCRIPTION:
The Study Drugs:

Methotrexate is designed to disrupt cells from making and repairing DNA (the genetic material of cells) and "copying" themselves.

Vincristine is designed to interfere with the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

Pegylated-L-asparaginase is designed to get rid of an important building block of proteins in leukemia cells.

Dexamethasone is a steroid that causes the leukemia cells to breakdown.

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive methotrexate through a needle in your vein on Days 1 and 15 (+/- 2 days) over 2 hours. You will receive vincristine by vein on Days 1, 8 and 15 (+/- 2 days) over 30 minutes. You will receive pegylated-L-asparaginase by vein on Days 2 and 16 (+/- 2 days) over about 2 hours. You will receive dexamethasone by vein over about 30 minutes or by mouth on Days 1-4 and 15-18 (+/- 2 days). If leukemia cells have a protein called cluster of differentiation antigen 20 (CD20), you will also receive rituximab by vein on Days 1 and 15 of Cycles 1-4 (+/- 2 days) over about 2-8 hours.

Each cycle will be at least 28 days.

If you have Philadelphia positive ALL, you may continue to receive a tyrosine kinase inhibitor (TKI). Examples of TKIs include Imatinib, Dasatinib, and Nilotinib. If you are not taking a TKI, you may begin taking a TKI. Your doctor will describe treatment with TKIs with you in more detail.

Once your blood counts improve and your leukemia is under control your doctor may decide to continue on treatment every 4-6 weeks. If your leukemia is not under control after the first cycle, your doctor may decide to start the next cycle without your blood counts improving.

Study Visits:

During Cycle 1, blood (about 2 teaspoons) will be drawn at least 1 time each week for routine tests. If the doctor thinks it is necessary, you may be asked to have additional blood drawn.

Between Days 14-28 of Cycle 1, you will have a bone marrow aspirate to check the status of the disease. This test may be delayed or repeated if your doctor does not think you are in remission.

Since pegylated-L-asparaginase can cause problems with blood clotting and inflammation of the pancreas, on Days 2 and 16 of All cycles, blood (about 2 teaspoons) will be drawn to check how well your blood clots and to check the health of your pancreas.

During Cycles 2- 6, blood (about 2 teaspoons) will be drawn for routine tests at least 2 times each month.

If the doctor thinks it is necessary, you may have a bone marrow aspirate to check the status of the disease.

Length of Study:

You may receive the study drugs for up to 6 cycles. You will be taken off study early if the disease gets worse, you experience intolerable side effects, or your doctor thinks that it is no longer in your best interest to receive the study drug(s).

This is an investigational study. Methotrexate, pegylated-L-asparaginase, and vincristine are all FDA approved for use in ALL. Dexamethasone is FDA approved as a steroid and steroids are traditionally an important part of treatment of leukemia. Rituximab is FDA approved for the treatment of non-Hodgkin's lymphoma. The combination of all these drugs is investigational.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Previously treated ALL (including Burkitt's lymphoma) or lymphoblastic lymphoma in relapse or primary refractory; without viable stem cell transplant option. Patients with previously treated Philadelphia chromosome positive ALL will be also eligible;
2. Chronic myeloid leukemia in blast phase
3. Zubrod performance status </= 3;
4. Adequate liver function (bilirubin </= 3.0mg/dl, unless considered due to tumor),and renal function (creatinine </= 3.0 mg/dl unless considered due to tumor;
5. Age >/= to 1 year
6. Understand and voluntarily sign an informed consent form.
7. For pediatric patients (age >/= 1 year to </= 18 years), Lansky performance status >/=50
8. For pediatric patients (age >/= 1 year to </= 18 years), second or greater relapse

Exclusion Criteria:

1. Pregnant patients
2. Prior history of allergic reaction, serious pancreatitis, hemorrhagic or thrombotic event with PEG-l-asparaginase or its components.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 6, 2009 to May 6, 2013. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Groups:
- MOAD: Chemotherapy regimen of methotrexate, rituximab, vincristine, pegylated L-asparaginase and dexamethasone (MOAD). Methotrexate 200 mg/m^2 intravenous (IV) days 1 and 15, Vincristine 1.4 mg/m^2 IV days 1, 8 and 15; PEG-l-asparaginase 2500 International units/m^2 IV days 2 and 16; Dexamethasone 40 mg/day IV or oral days 1-4 & 15-18; Rituximab 375 mg/m^2 IV days 1 & 15 (first 4 cycles) for participants CD20 positive or positive by immunostain.
Period: Overall Study
Arm/Group | MOAD
Started | 37
Completed | 36
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | MOAD
Number analyzed (Participants) | 37
Age, Continuous [Mean (Full Range); unit: years] | 42 [22 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate
Description: Rate calculated as number of participants with CR. Complete Remission (CR) defined as Normalization of peripheral blood and bone marrow with 5% or less blasts in a normocellular or hypercellular marrow with a granulocyte count of 1 x 10^9/L or above and platelet count of 100 x 10^9/L or above. Complete resolution of all sites of extramedullary disease is required for CR.
Time Frame: 6 cycles (cycle = 28 days)
Population: Of the 37 participants enrolled, 36 participants completed therapy and were evaluable for response.
Measure: Number; unit: percentage of participants
Arm/Group | MOAD
Number analyzed (Participants) | 36
percentage of participants | 28

ADVERSE EVENTS:
Time Frame: Adverse events collected through 28 day cycle, up to six cycles. Overall collection period: April 2009 to February 2013.
Description: The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | MOAD
Serious Adverse Events (participants affected / at risk) | 33/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOAD (N=37)
Cardiopulmonary Arrest (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 4 (5)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 4 (4)
Nausea and Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal Pain (General disorders) | 1 (1)
Death (General disorders) | 14 (14)
Weakness (General disorders) | 3 (3)
Hepatic Abcess (Hepatobiliary disorders) | 1 (1)
Liver Dysfunction (Hepatobiliary disorders) | 1 (1)
Liver Failure (Hepatobiliary disorders) | 2 (2)
Bacteremia (Infections and infestations) | 1 (1)
Candida Gabrata Infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Colitis (Infections and infestations) | 1 (1)
Infection due to Catheter (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (2)
Neutropenic Fever (Infections and infestations) | 7 (8)
Osteomyelitis (Infections and infestations) | 1 (1)
Pancreatitis (Infections and infestations) | 2 (2)
Parotiditis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 9 (9)
Sepsis (Infections and infestations) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Septicemia (Infections and infestations) | 1 (1)
Elevated Alanine transaminase (Metabolism and nutrition disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Right Hip Fracture/Fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Altered Mental Status (Nervous system disorders) | 2 (2)
Paralysis due to CNS disease (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Leptomeningeal disease (Eye disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOAD (N=37)
Elevated Liver Enzymes (Hepatobiliary disorders) | 34 (34)
Elevated bilirubin (Hepatobiliary disorders) | 31 (31)
Decreased fibrinogen (Blood and lymphatic system disorders) | 26 (26)
Nausea (Gastrointestinal disorders) | 11 (11)
Neuropathy (Nervous system disorders) | 10 (10)
Elevated amylase/lipase (Metabolism and nutrition disorders) | 9 (9)
Mucositis (Gastrointestinal disorders) | 8 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Thrombosis (Vascular disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (4)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Infection (Infections and infestations) | 26 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes